CLINICAL TRIAL: NCT04614155
Title: Texas State HPV Self-Collection Pilot Study
Brief Title: Project Self in Improving Cervical Cancer Screening Rates in Hispanic and African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-0182; NCI-2019-04860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0182 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-26; First posted 2020-11-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (questionnaire, health education, self-collection) (Experimental): Participants complete questionnaires, take part in a health education session, and receive HPV self-collection kit.
  Interventions: Other: Educational Intervention; Procedure: HPV Self-Collection; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Take part in health education session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Procedure: HPV Self-Collection — Receive HPV self-collection kit
  Other Names: At-home HPV Self Collection; HPV Self Collection; Human Papillomavirus Self-Collection
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial studies if Project Self can improve the rate of cervical cancer screening in Hispanic and African American women living in Houston, Texas. Project Self may help to improve cervical cancer screening rates by providing human papillomavirus (HPV) self-collection kits, education, counseling, and navigation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the feasibility of conducting an education intervention trial regarding cervical cancer screening among women of Hispanic and African American origin living in public housing units in Houston, Texas.

SECONDARY OBJECTIVES:

I. Document cervical screening associated knowledge, attitudes and practices among Hispanic and African American women living in public housing units in Houston, Texas at pre- and post-health education.

II. Document Pap smear screening rate in last 3 years among participants. III. Document HPV positive rate among participants.

OUTLINE:

Participants complete questionnaires, take part in a health education session, and receive an HPV self-collection kit.

After completion of study, participants are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American or Hispanic women.
* Valid home address reflective of residence in the participating housing development(s) at least 50% of the time.
* Functioning telephone number.
* Speak and read English or Spanish.

Exclusion Criteria:

* Self-reported hysterectomy.
* Self-reported personal history of cancer/cancer diagnosis.
* Self-reported as pregnant.
* Another household member is enrolled in this protocol.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Participant consent rate | Up to 1 month
Human papillomavirus (HPV) self-collection uptake rate | Up to 2 weeks after health education session
  Defined as the proportion of the participants who consent to the study and receive an HPV self-collection kit complete the self-collection and return the sample to the lab or research staff member or community health worker within timeline.

SECONDARY OUTCOMES:
Cervical screening associated knowledge, attitudes and practices score | Up to 1 month
  Paired t-tests or Wilcoxon signed-rank tests will be used to examine the change of the scores difference for cervical screening associated knowledge, attitudes and practices. For every participant, 'Knowledge' will be measured using a 12-question scale, which will have a 'Yes/No/Unsure' response. Each 'correct' response will be scored as 1, while 'incorrect' and 'unsure' as 0. A score 50% (≥6 correct responses) will be considered as optimal. 'Attitude' will be measured using a 6-question scale which will have 'Disagree/Neutral/Agree response. Attitude will be considered as favorable if we have three or more "Agree" responses. Being screened, before our education-intervention, for cervical cancer with Pap-smear, and after our intervention either with HPV self-sampling or Pap-smear, will be regarded as having good practice. Changes in Knowledge, Attitude and Practice, pre- and post-education intervention will be examined using Paired t-tests or Wilcoxon signed-rank tests.
Participants' self-reported Pap smear screening rate in last 3 years | Up to 1 month
HPV positive proportion | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Surendranath S Shastri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shastri SS, McNeill LH, Shete S. Culturally Competent Education and Human Papillomavirus Self-Sampling Achieves Healthy People 2030 Cervical Screening Target Among Low-Income Non-Hispanic Black and Hispanic Women. JCO Glob Oncol. 2024 May;10:e2400005. doi: 10.1200/GO.24.00005. PMID 38723214
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT04614155/ICF_000.pdf